CLINICAL TRIAL: NCT03891290
Title: Collecting Recorded Videos of Colonoscopy Screening Tests for the Evaluation of the Automatic Polyp Detection System (APDS) Medical Device
Brief Title: Collecting Recorded Videos of Colonoscopy Screening Tests
Status: Completed | Type: Observational
Sponsor: Magentiq Eye LTD (Industry)
Responsible Party: Sponsor
Other Study IDs: 0009-16-HYMC
Record Dates: First submitted 2019-03-09; First posted 2019-03-27 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Colon Polyp
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Collecting recorded videos of Colonoscopy screening tests of the general population — To evaluate, in objective way, the usability of the future alpha version of the APDS device by testing the sensitivity and specificity of its results achieved from running it on the collected recorded videos of Colonoscopy screening tests of the general population.

SUMMARY:
The study shall mainly help to better evaluate the performance the APDS device and secondly it may help to assess the potential of the future alpha version of the device to be a useful and effective for the detection of colon Polyps.

DETAILED DESCRIPTION:
Primary objectives • To evaluate, in objective way, the usability of the future alpha version of the APDS device by testing the sensitivity and specificity of its results achieved from running it on the collected recorded videos of Colonoscopy screening tests of the general population.

Secondary objectives

• When the APDS would be ready for field installation (Beta Version), to install it in the Gastroenterology institute of the medical center, in order to evaluate, as part of a continuation study, the physicians satisfaction from the APDS performance.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all the criteria related to regular colonoscopy according to the standard of care at the Gastroenterolgy Department of the selected center. In addation, the following criteria have to be met to be eligible for the study:

1. Able to read, understand and provide written Informed Consent;
2. Females or males - older than 18 years old

Exclusion Criteria:

Any of the following colonoscopy related exclusion criteria will exclude the subject from the study:

* Bleeding disorder or unacceptable risk of bleeding
* Terminal illness or life threatening malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects shall be recruited by the investigator from within the investigator's patient population of colonoscopy. In this study one site will participate and enroll up to 300 subjects according to the inclusion/exclusion criteria. Each subject (up to 300 subjects) included will pass one regular colonoscopy screening test which will be recorded in the way which is described above.
  Enrolled subjects that did not complete the full course of the study will be replaced.
Sampling Method: Non-Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2016-11-21 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2019-07-10 (Actual)

PRIMARY OUTCOMES:
Recorded colonoscopy video which was verified by visual inspection to have sufficient high quality. | Half an hour from the end of the procedure at which the video was recorded.
  Each recorded video is visually inspected immediately at the end of the procedure by an experienced team member who rates it with a number between 1 (low quality) to 10 (high quality). Only videos with rate above 7 are considered as having sufficient high quality.
De-Identified procedure report which was visually inspected to verify that it includes all the needed details about the polyps that were detected during the procedure. | Half an hour from the end of the procedure for which the procedure report was filled-in.
  Each de-Identified procedure report is visually inspected immediately at the end of the procedure by an experienced team member who gives it binary score (0 or 1), 1 if it includes all the needed details about the polyps that were detected during the procedure, and 0 if it does not include all the needed details about the polyps that were detected during the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Yael Kopelman, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No